CLINICAL TRIAL: NCT03745313
Title: Edwards PASCAL TrAnScatheter Valve RePair System in Tricuspid Regurgitation (CLASP TR) Early Feasibility Study
Brief Title: Edwards CLASP TR EFS
Acronym: CLASP TR EFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Tricuspid Regurgitation
Keywords: Functional; TR; FTR; Transcatheter; Repair; Regurgitation; Degenerative
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the Edwards PASCAL Transcatheter Valve Repair System
  Interventions: Device: Edwards PASCAL Transcatheter Valve Repair System

INTERVENTIONS:
Device: Edwards PASCAL Transcatheter Valve Repair System — Repair of the tricuspid valve through a transcatheter approach

SUMMARY:
Early feasibility study to assess the safety and performance of the Edwards PASCAL Transcatheter Valve Repair System in tricuspid regurgitation

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-arm, and non-randomized study designed to evaluate the safety and performance of the Edwards PASCAL Transcatheter Valve Repair System

ELIGIBILITY:
Inclusion Criteria:

* Severe functional or degenerative TR
* Symptomatic despite medical therapy
* The local site Heart Team determines that the patient is appropriate for transcatheter tricuspid valve repair

Exclusion Criteria:

* Unsuitable anatomy
* Previous tricuspid valve repair or replacement
* Co-morbid condition(s) that, in the opinion of the investigator, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2025-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susheel K. Kodali, MD, Principal Investigator — Columbia University
Locations (15):
- United States (15):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kodali SK, Hahn RT, Davidson CJ, Narang A, Greenbaum A, Gleason P, Kapadia S, Miyasaka R, Zahr F, Chadderdon S, Smith RL, Grayburn P, Kipperman RM, Marcoff L, Whisenant B, Gonzales M, Makkar R, Makar M, O'Neill W, Wang DD, Gray WA, Abramson S, Hermiller J, Mitchel L, Lim DS, Fowler D, Williams M, Pislaru SV, Dahou A, Mack MJ, Leon MB, Eleid MF. 1-Year Outcomes of Transcatheter Tricuspid Valve Repair. J Am Coll Cardiol. 2023 May 9;81(18):1766-1776. doi: 10.1016/j.jacc.2023.02.049. PMID 37137586
- [Derived] Kodali S, Hahn RT, Eleid MF, Kipperman R, Smith R, Lim DS, Gray WA, Narang A, Pislaru SV, Koulogiannis K, Grayburn P, Fowler D, Hawthorne K, Dahou A, Deo SH, Vandrangi P, Deuschl F, Mack MJ, Leon MB, Feldman T, Davidson CJ; CLASP TR EFS Investigators. Feasibility Study of the Transcatheter Valve Repair System for Severe Tricuspid Regurgitation. J Am Coll Cardiol. 2021 Feb 2;77(4):345-356. doi: 10.1016/j.jacc.2020.11.047. PMID 33509390

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards PASCAL Transcatheter Tricuspid Valve Repair System: Tricuspid valve repair with PASCAL implanted via transcatheter procedure
Period: At 30 Days Follow-up
Arm/Group | Edwards PASCAL Transcatheter Tricuspid Valve Repair System
Started | 65
Completed | 63
Not Completed | 2
Not completed — Death | 2
Period: At 6 Months Follow-up
Arm/Group | Edwards PASCAL Transcatheter Tricuspid Valve Repair System
Started | 57
Completed | 54
Not Completed | 3
Not completed — Death | 1
Not completed — Missed Visit | 1
Not completed — Exited for Other Reason Within Window | 1
Period: At 1 Year Follow-up
Arm/Group | Edwards PASCAL Transcatheter Tricuspid Valve Repair System
Started | 51
Completed | 47
Not Completed | 4
Not completed — Death | 2
Not completed — Missed Visit | 2
Period: At 2 Year Follow-up
Arm/Group | Edwards PASCAL Transcatheter Tricuspid Valve Repair System
Started | 43
Completed | 42
Not Completed | 1
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants who received any amount of study drug
Arm/Group | Edwards PASCAL Transcatheter Tricuspid Valve Repair System
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.4 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: Kilogram Per Meter Squared] — Population: Data unavailable for 2 patients.
  Kilogram Per Meter Squared
    number analyzed (Participants) | 63
    (all) | 26.7 (5.81)
Tobacco Use [Count of Participants; unit: Participants]
  Current Daily Smoker | 0
  Former Daily Smoker | 26
  Never | 39
NYHA Class [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    Class I | 1
    Class II | 18
    Class III | 44
    Class IV | 2
EuroSCORE II [Mean (Standard Deviation); unit: Units on a scale] — EuroScore II is a risk model which allows the calculation of the risk of death after a heart operation. Scores range from a minimum of 0 to a maximum of 100.
  EuroScore II risk levels are as follows:
  < 8: Low risk; 8-10: Moderate risk; >10: High risk Population: Data unavailable for 3 patients.
  Units on a scale
    number analyzed (Participants) | 62
    (all) | 5.0 (4.69)
STS Mortality Score [Mean (Standard Deviation); unit: Units on a scale] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. Scores range from a minimum of 0 to a maximum of 100. An STS predicted risk of surgical mortality of 4-8 is considered intermediate risk; and a score 8 or greater is considered high risk. The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator calculates a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries. Population: Data unavailable for 1 patient.
  Units on a scale
    number analyzed (Participants) | 64
    (all) | 7.4 (5.21)
Clinical Frailty Total Score [Count of Participants; unit: Participants]
  Non-Frail | 50
  Mild-to-Moderately Frail | 15
  Severely Frail | 0
Katz Activities of Daily Living Total Score [Mean (Standard Deviation); unit: Units on a scale] — The Katz Activities of Daily Living (ADL) scale is a widely used graded instrument that assesses six primary and psychosocial functions: bathing, dressing, going to toilet, transferring, feeding, and continence.
  Scoring:
  6 = High (patient independent). 4 = Moderate (patient is moderately functioning). 0-2 = Low (patient very dependent).
  Units on a scale | 5.8 (0.48)
Modified Rankin Scale [Count of Participants; unit: Participants] — Population: Data unavailable for 59 patients.
  Participants
    number analyzed (Participants) | 6
    No symptoms at all | 3
    No significant disability despite symptoms | 2
    Moderate disability | 1

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Event (MAE) Rate
Description: Number and percentage of patients who experienced at least one major adverse event (MAE). Composite of major adverse events (MAE) defined as cardiovascular mortality, myocardial infarction (MI), stroke, renal complications requiring unplanned dialysis or renal replacement therapy, severe bleeding, unplanned or emergency re-intervention related to the device, and major access site and vascular complications requiring intervention at 30 days.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Valve Repair System
Number analyzed (Participants) | 65
Participants | 6

2. Secondary Outcome: Device Success
Description: Number and percentage of Device Success, definition modified from MVARC criteria. Per device analysis
Time Frame: Intraprocedural
Population: Per device analysis
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Edwards PASCAL Transcatheter Valve Repair System
Number analyzed (Participants) | 65
Number analyzed (Device) | 103
Device | 90

3. Secondary Outcome: Procedural Success
Description: Number and percentage of patients who had Procedural Success, definition modified from MVARC criteria. Per patient analysis
Time Frame: Discharge (2-7 days)
Population: The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Valve Repair System
Number analyzed (Participants) | 56
Participants | 49

4. Secondary Outcome: Clinical Success
Description: Number and percentage of patients who had procedural success without MAEs at 30 days. Per patient analysis
Time Frame: 30 days
Population: The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Valve Repair System
Number analyzed (Participants) | 56
Participants | 43

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Edwards PASCAL Transcatheter Valve Repair System
All-Cause Mortality (participants affected / at risk) | 24/65
Serious Adverse Events (participants affected / at risk) | 49/65
Other Adverse Events (participants affected / at risk) | 57/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards PASCAL Transcatheter Valve Repair System (N=65)
Anaemia (Blood and lymphatic system disorders) | 5 (7)
Atrial Fibrillation (Cardiac disorders) | 4 (6)
Cardiac Failure (Cardiac disorders) | 8 (13)
Cardiac Failure Congestive (Cardiac disorders) | 10 (14)
Tricuspid Valve Incompetence (Cardiac disorders) | 5 (5)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 (4)
Death (General disorders) | 5 (5)
Pneumonia (Infections and infestations) | 5 (6)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 13 (18)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 9 (12)
Cerebrovascular Accident (Nervous system disorders) | 4 (4)
Acute Kidney Injury (Renal and urinary disorders) | 8 (10)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Vascular Disorders (Vascular disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards PASCAL Transcatheter Valve Repair System (N=65)
Tricuspid Valve Incompetence (Cardiac disorders) | 13 (13)
Cardiac Failure Congestive (Cardiac disorders) | 11 (15)
Atrial Fibrillation (Cardiac disorders) | 7 (9)
Cardiac Failure Acute (Cardiac disorders) | 5 (5)
COVID-19 (Infections and infestations) | 6 (6)
Pneumonia (Infections and infestations) | 6 (8)
Urinary Tract Infection (Infections and infestations) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 9 (9)
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Syncope (Nervous system disorders) | 6 (7)
Cerebrovascular Accident (Nervous system disorders) | 4 (4)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 (5)
Acute Kidney Injury (Renal and urinary disorders) | 15 (18)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (7)
Hypotension (Vascular disorders) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 7 (9)
Investigations (Investigations) | 8 (9)
Psychiatric Disorders (Psychiatric disorders) | 4 (5)
Surgical and Medical Procedures (Surgical and medical procedures) | 4 (4)
Cardiac Failure (Cardiac disorders) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03745313/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03745313/SAP_003.pdf